CLINICAL TRIAL: NCT02879968
Title: Correlation Between Serum Squamous Cell Carcinoma Antigen Level and Tumor Volume in Head and Neck Cancer
Brief Title: Serum Squamous Cell Carcinoma Antigen Level and Tumor Volume in Head and Neck Cancer
Status: Completed | Type: Observational
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Kitti Jantharapattana, M.D., Assistant Professor, Prince of Songkla University
Other Study IDs: PrinceSongklaU
Record Dates: First submitted 2016-08-23; First posted 2016-08-26 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Head and Neck Cancer
Keywords: serum squamous cell carcinoma antigen; tumor volume; Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum squamous cell carcinoma antigen
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Head and Neck squamous cell carcinoma: A single measurement of serum squamous cell carcinoma antigen level is performed in the eligible Head and Neck squamous cell carcinoma patients.
  The study tool measuring serum squamous cell carcinoma antigen level is ARCHITECT SCC (Abbott).
  The gross tumor volume in the cross sectional imaging obtained within 2 weeks of each patient is calculated with the typical ellipsoid formula.
  Interventions: Other: Non-interventional study

INTERVENTIONS:
Other: Non-interventional study

SUMMARY:
Correlation between serum squamous cell carcinoma antigen level and tumor volume in Head and Neck Cancer is to determine a correlation between level of serum squamous cell carcinoma antigen and tumor volume in Head and Neck Caner measured by cross-sectional imaging.

DETAILED DESCRIPTION:
The study is a cross-sectional study. A single measurement of serum squamous cell carcinoma antigen level is performed in the eligible Head and Neck squamous cell carcinoma patients.

The study tool measuring serum squamous cell carcinoma antigen level is ARCHITECT SCC (Abbott).

The gross tumor volume in the cross sectional imaging obtained within 2 weeks of each patient is calculated with the typical ellipsoid formula.

Correlation between both parameters will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven squamous cell carcinoma in Head and Neck
* Getting a cross-sectional imaging of Head and Neck within 2 weeks of collecting serum squamous cell carcinoma antigen

Exclusion Criteria:

* Metastatic disease
* Accompanied Non-Head and Neck squamous cell carcinoma
* Nasopharyngeal, thyroid, salivary, nose and paranasal sinus carcinoma
* Skin disease: eczema, erythrodermic epidermitis, pemphigus, and psoriasis
* Pulmonary disease: tuberculosis, adult respiratory distress syndrome, pulmonary infiltration with eosinophilia, sarcoidosis, and bronchogenic cyst
* Renal failure
* Using antihistamine eye drops

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Head and Neck squamous cell carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2016-08; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Correlation between serum squamous cell carcinoma antigen and tumor volume | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Prince of Songkla University, Hadyai, Changwat Songkhla, Thailand

IPD SHARING:
Plan to Share IPD: No